CLINICAL TRIAL: NCT06126029
Title: Effect of Metformin as Add-on Therapy to Ibuprofen on Disease Activity in Knee Osteoarthritis Patients: A Randomized Controlled Trial.
Brief Title: Effect of Metformin as Add-on Therapy to Ibuprofen on Disease Activity in Knee Osteoarthritis Patients.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Delowar Hossain, MD, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BSMMU/2023/11020
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Knee Osteoarthritis; Metformin
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin group (Experimental): This group will receive metformin 500mg extended release oral tablet daily along with standard of care for 8 weeks.
  Interventions: Drug: Metformin 500 Mg extended release Oral Tablet
- Placebo group (Placebo Comparator): This group will receive placebo oral tablet daily along with standard of care for 8 weeks.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Metformin 500 Mg extended release Oral Tablet — 34 patients of experimental group will get metformin 500mg extended release oral tablet once daily with evening meal along with standard of care (ibuprofen 400mg and rabeprazole 20mg twice daily) for 8 weeks as prescribed by the physician.
  Arms: Metformin group
Drug: Placebo oral tablet — 34 patients of placebo group will get placebo oral tablet once daily with evening meal along with standard of care (ibuprofen 400mg and rabeprazole 20mg twice daily) for 8 weeks as prescribed by the physician.
  Arms: Placebo group

SUMMARY:
The goal of this randomized, double blind, placebo-controlled clinical trial is to learn about, the effect of metformin compared with placebo-controlled group on disease activity and interleukin-6 level in patients with knee osteoarthritis.The main question it aims to answer is:Is Metformin as add-on therapy more effective in reducing disease activity in Ibuprofen-treated patients with grade II-III knee osteoarthritis? Half of Participants will receive metformin with standard of care(ibuprofen and rabeprazole) while other half placebo and standard of care (ibuprofen and rabeprazole).

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a worldwide highly prevalent chronic joint disease commonly affecting individuals of 40 years and older. OA is highly debilitating, encompassing various physical symptoms like pain, stiffness, swelling, disability and loss of normal joint function. Knee OA is one of the major causes of impaired function and disability of elderly population resulting in markedly reduced quality of life and increased socioeconomic burden.

(OA) is a progressive degenerative disorder characterized by degraded cartilage,low to moderate synovial inflammation, alteration of bony structure.The pathogenesis of OA is complex, combination of risk factors such as aging, obesity, being female, smoking, genetics, excessive joint load and injury, metabolic alterations and mechanical stress contribute to OA.These factors induce low-grade chronic inflammation and imbalance in oxidant-antioxidant levels, stimulating chondrocytes to produce reactive oxygen species (ROS) and pro-inflammatory cytokines. Overproduction of IL-1β, IL-6, TNF-α activate synoviocytes,macrophages, B and T lymphocytes, chondrocytes to play a role in the cartilage degradation, a central feature of OA.The infrapatellar fat pad (IFP) from knee OA patients secreted significantly higher levels of IL-6, but not TNF-α and IL-1β.

Decreased AMPK-α activity was found in human samples as well as mice OA knee joint chondrocytes which leads to increased mTOR activity,inhibition of autophagy, increased apoptosis and inflammatory activity of OA chondrocytes. Mitochondrial injury and a lowered expression of SIRT1 protein are often associated with the pathogenesis of OA.

Existing therapies such as Nonsteroidal Anti-inflammatory drugs (NSAIDs) and other analgesics are only used to reduce pain and swelling. With the chronic nature of knee OA, pharmacological approaches must be safe for long-term use. NSAIDs are the mainstay of management for knee OA but cause serious gastrointestinal, renal and cardiovascular adverse events with no beneficial effect on joint structures.Total knee replacement is the last option for patients with end-stage knee OA.

Metformin exerts a chondroprotective effect by inducing the SIRT1 expression and activating AMPK-α, leading to reduced inflammatory mediators and matrix degradation substances, inhibit the accumulation of RAGE, increase in autophagy as well as a decrease in catabolism and apoptosis, as evidenced by in vivo and in vitro studies. Metformin as an AMPK-α activator can protect inflammatory cell death of chondrocytes and attenuates cartilage degeneration and prevents or delays the development and progression of knee OA. Metformin is able to reduce RANKL and stimulates OPG expression in osteoblasts, further inhibit osteoclast differentiation and prevent bone loss. Data from human studies suggest that metformin could reduce knee OA progression by modifying inflammatory pathways and being considered as an alternative or adjuvant treatment of knee OA.

This study is a double-blind, randomized, placebo-controlled trial in knee OA patients. This study will be conducted to evaluate the effect of metformin as add-on therapy on disease progression and inflammatory indicator in knee OA patients.The intervention group will receive metformin 500mg extended release tablet once daily for 8 weeks, with standard of care(ibuprofen and rabeprazole) as prescribed by the physician whereas control group will receive placebo oral tablet once daily with standard of care(ibuprofen and rabeprazole) during the same study period. The investigator will compare changes in five dimensions (pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life) of KOOS score (out of 100) and serum interleukin-6 (IL-6) level, at the time of recruitment with after 8 weeks of intervention in both the intervention and placebo controlled groups.

Adding Metformin with the conventional treatment of Ibuprofen could potentially have a substantial impact on disease activity in patients with Knee Osteoarthritis(OA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee pain
* Radiographic evidence of knee osteoarthritis (Grade II-III)
* Age 18-65 years
* Both male and female
* Normal BMI(for asians): 18.5-22.9 kg/m2

Exclusion Criteria:

* Diagnosed case of Diabetes Mellitus, renal, hepatic, cardiovascular or pulmonary disease
* Diagnosed case of Gout or pseudogout
* Diagnosed case of systemic inflammatory conditions such as rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease
* Patients currently receiving immunosuppressant, carbonic anhydrase inhibitors(topiramate), ranolazine, vandetanib, dolutegravir
* History of receiving a corticosteroid injection in the last three months
* Prior history of knee trauma or surgery
* Metformin use or history of use in the last two months
* Known allergy to metformin
* History of lactic acidosis
* Patient with habit of excessive alcohol intake
* Pregnancy
* Patients unwilling to participate or unwilling to give written consent
* Participation in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 1 year
  The KOOS meets basic criteria of outcome measures and can be used to evaluate the course of knee injury and treatment outcome. KOOS will be used to assess improvements in the scores(out of 100) of five patient-relevant outcomes (pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life) of knee osteoarthritis patients after 8 weeks of intervention.

SECONDARY OUTCOMES:
Serum Interleukin-6 (IL-6) level | 1 year
  The reported values for IL-6 in the blood of healthy donors varied between 0 and 43.5 pg/ml.The pooled estimate of IL-6 was 5.186 pg/ml. IL-6 follows a circadian rhythm with a peak at the time of waking (04 am).Significantly higher levels of IL-6 are secreted from the Infrapatellar fat pad of knee OA patients and correlate with disease progression or severity of cartilage pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Md.Delowar Hossain, MD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes